CLINICAL TRIAL: NCT07219316
Title: Regenerative High Purity Type I Collagen Scaffold for Breast Volume Restoration Following Breast-Conserving Surgery: A Multicentre Prospective Clinical Trial
Brief Title: Regenerative Collagen Scaffold for Breast Volume Restoration in Breast-Conserving Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adichunchanagiri Institute of Medical Sciences, B G Nagara (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIMS/IEC/240/2025
Record Dates: First submitted 2025-10-17; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Breast-Conserving Surgery
Keywords: Breast-Conserving Surgery; Volume Restoration; Collagen Matrix; Breast Reconstruction; Regenerative Scaffold; High Purity Type I Collagen; Oncoplastic Surgery; Surgicoll-Mesh

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- High Purity Type I Collagen Scaffold (Experimental): Patients undergoing breast conservative surgery will receive immediate placement of high purity Type I collagen scaffold to fill tissue defect. The scaffold is a sterile, cross-linked bovine Type I collagen matrix with degradation time of 2 months, sterilized by ethylene oxide
  Interventions: Device: High Purity Type I Collagen Scaffold (Regenerative Matrix)

INTERVENTIONS:
Device: High Purity Type I Collagen Scaffold (Regenerative Matrix) — Standard breast-conserving surgery followed by immediate scaffold placement into the excision cavity. The scaffold is sutured using absorbable sutures and covered with standard wound closure. Postoperative care follows institutional protocols. Adjuvant radiotherapy and chemotherapy as indicated per oncological protocols; standard antibiotics and analgesics.

SUMMARY:
This clinical trial evaluates the safety and efficacy of High Purity Type I Collagen scaffold for breast volume restoration following breast-conserving surgery (BCS). The regenerative collagen matrix serves as a biocompatible scaffold promoting tissue ingrowth, neovascularization, and gradual remodeling, thereby improving cosmetic outcomes and patient quality of life after partial mastectomy.

DETAILED DESCRIPTION:
Breast-conserving surgery (BCS) is the standard treatment for early-stage breast cancer, balancing oncological safety with aesthetic preservation. However, postoperative volume defects may cause breast asymmetry and psychological distress. Traditional options such as flaps or implants are limited by donor-site morbidity and complications.

This prospective, single-arm, bi-centre study investigates the clinical performance of a high-purity, cross-linked bovine Type I collagen scaffold for immediate breast volume restoration. The study will assess safety, volume maintenance, cosmetic appearance, and patient-reported outcomes through standardized 3D imaging, MRI analysis, and validated quality-of-life instruments.

The study will enroll 40 women undergoing BCS with expected volume defects ≥20%, with 2-month postoperative follow-up for primary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18-70 years
* Histologically confirmed breast carcinoma (Stage 0-II) or high-risk lesions requiring excision
* Expected postoperative defect ≥20% of total breast volume
* ECOG 0-1, adequate organ function
* Informed consent provided, compliant with follow-up schedule

Exclusion Criteria:

* Prior breast surgery or radiotherapy to affected breast
* Locally advanced or inflammatory carcinoma
* Collagen hypersensitivity or autoimmune disease
* Active infection, pregnancy, lactation, or smoking within 6 weeks
* Concurrent participation in other clinical studies

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Volume restoration | 2 months post-operative
  Proportion of patients achieving ≥80% breast volume retention at 2 months assessed by imaging/MRI
Patient satisfaction with breast volume restoration | 2 months post-operative
  Patient satisfaction ≥7/10 on standardized satisfaction scale (BREAST-Q). The BREAST-Q is a validated patient-reported outcome measure (PROM) used to assess the quality of life and satisfaction of patients undergoing breast surgery. It consists of specific modules for different procedures, like reconstruction, and measures aspects such as psychological well-being, physical well-being (chest and sexual), and satisfaction with the breasts and care. The scale, which results in scores from 0 to 100, helps evaluate the impact of surgery from the patient's perspective. Scores range from 0 to 100, with higher scores indicating a greater degree of health-related quality of life or satisfaction.

SECONDARY OUTCOMES:
Objective Volume Assessment | 2 months post-operative
  Percentage change in breast volume at 2, 4, and 8 weeks post-surgery
Breast Volume symmetry index | 2 months post-operative
  Volume symmetry index - operated vs. contralateral breast. The Breast Volume Symmetry Index (BVSI) quantifies postoperative symmetry between the operated and contralateral (unoperated) breasts. It is calculated as the ratio of the breast volume on the operated side to that of the contralateral side, multiplied by 100 to express as a percentage:
  BVSI = (Operated Breast Volume / Contralateral Breast Volume) × 100. A value of 100% indicates perfect symmetry, while lower values indicate volume deficit.
Cosmetic Assessment | 2 months post-operative
  Physician-rated 4-point cosmetic score. This is a standardized visual assessment tool used to evaluate the aesthetic outcome of the operated breast compared to the contralateral breast. The assessment is based on parameters such as breast shape, volume, symmetry, contour, nipple-areolar complex position, and scar appearance. The 4-point grading system is typically defined as:
  Grade 4 - Excellent - Described as operated breast almost identical to contralateral side - Criteria is minimal asymmetry, natural contour Grade 3 - Good - Described as slight difference in shape or volume - Acceptable symmetry and cosmetic result Grade 2 - Fair - Described as noticeable asymmetry or distortion - Moderate contour irregularity or scar visibility Grade 1 - Poor - Described as significant deformity or volume loss - Unacceptable cosmetic result
Radiological Outcomes | 2 months
  MRI Scoring System - Scaffold Integration, Vascularization & Resorption:
  Standardized MRI assessment of scaffold performance (integration, neovascularization, resorption) at baseline, Week 4, and Week 8.
  MRI protocol:
  T1 (axial/sagittal), T2/STIR (axial), DCE T1 (pre-contrast, early 30-60 s, intermediate 90-120 s, delayed 4-6 min),
  Scores (0-3 each):
  A. Integration: 0 = none; 1 = minimal; 2 = moderate; 3 = complete tissue continuity.
  B. Vascularization: 0 = none; 1 = mild/delayed; 2 = moderate (neovascular); 3 = marked (early enhancement).
  C. Resorption: 0 > 75% residual; 1 = 50-75%; 2 = 25-50%; 3 < 25% residual. D. Tissue Quality: 0 = fluid-filled; 1 = mostly fluid; 2 = mixed; 3 = tissue-like.
  Composite MRI Integration Score (MIS 0-12): Higher = better integration/remodeling.
  Interpretation:
  0-3 Poor, 4-7 Moderate, 8-10 Good, 11-12 Excellent.
Complications | 2 months
  Incidence of seroma, hematoma, infection, abscess, wound dehiscence, or scaffold exposure / extrusion, suspicious lump requiring biopsy
Pain Assessment | 2 months
  Pain assessment at 1, 2, 4 and 8 weeks post surgery using Visual Analogue Scale (VAS). The VAS is a simple, validated tool used to measure the intensity of pain. It consists of a 10-centimeter horizontal line with two extreme anchors: 0 = No pain and 10 = Worst imaginable pain.
  Participants are asked to mark a point on the line that best represents their current perception of pain. The score is determined by measuring, in millimeters, the distance from the "0" end to the participant's mark. VAS provides a continuous, quantitative measure of subjective outcomes that is easy to administer, sensitive to small changes, and widely used in post-surgical pain assessment

CONTACTS AND LOCATIONS:
Overall Officials: Prema Dhanraj, MS, MCh, Study Chair — Rajarajeswari Medical College and Hospital
Locations (2):
- India (2):
  - Adichunchanagiri Institute of Medical Sciences, Mandya, Karnataka
  - JSS Medical College Hospital, Mysore, Karnataka

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets will be available upon reasonable request following publication of primary results.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months post-publication
Access Criteria: Researchers providing methodologically sound proposals with IRB approval

REFERENCES:
- [Background] Narayan N, Shivannaiah C, Gowda S. Evaluating the Efficacy of High-Purity Type I Collagen-Based Skin Substitute Versus Dehydrated Human Amnion/Chorion Membrane in the Treatment of Venous Leg Ulcers: A Randomized Controlled Clinical Trial. Cureus. 2025 Jul 30;17(7):e89031. doi: 10.7759/cureus.89031. eCollection 2025 Jul. PMID 40747200
- [Background] Narayan N, Gowda S, Shivannaiah C. A Randomized Controlled Clinical Trial Comparing the Use of High Purity Type-I Collagen-Based Skin Substitute vs. Dehydrated Human Amnion/Chorion Membrane in the Treatment of Diabetic Foot Ulcers. Cureus. 2024 Dec 5;16(12):e75182. doi: 10.7759/cureus.75182. eCollection 2024 Dec. PMID 39649230
- [Background] van Loevezijn AA, Geluk CS, van den Berg MJ, van Werkhoven ED, Vrancken Peeters MTFD, van Duijnhoven FH, Hoornweg MJ. Immediate or delayed oncoplastic surgery after breast conserving surgery at the Netherlands Cancer Institute: a cohort study of 251 cases. Breast Cancer Res Treat. 2023 Apr;198(2):295-307. doi: 10.1007/s10549-022-06841-8. Epub 2023 Jan 24. PMID 36690822
- [Background] Slavin SA, Halperin T. Reconstruction of the breast conservation deformity. Semin Plast Surg. 2004 May;18(2):89-96. doi: 10.1055/s-2004-829043. PMID 20574487
- [Background] Narayan N, Ramegowda YH, Raghupathi DS, Chethan S, Gowda S. Biological Skin Substitutes in Pressure Ulcers: High-Purity Type I Collagen-Based Versus Amnion/Chorion Membrane. Cureus. 2025 Aug 25;17(8):e90956. doi: 10.7759/cureus.90956. eCollection 2025 Aug. PMID 40862036